CLINICAL TRIAL: NCT06249659
Title: Impact of Extubation Location After Surgery on Perioperative Times. A Prospective Multicenter Observational Study. Extub_Loca Study
Brief Title: Impact of Extubation Location After Surgery on Perioperative Times
Acronym: Extub_Loca
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-MTP_2022_04_202201100
Record Dates: First submitted 2024-01-04; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Anesthesia; Intubation; Surgery; Extubation; Respiratory Failure; Complication,Postoperative
Keywords: General anesthesia; Extubation; Intubation; Time; Complications
MeSH Terms: conditions — Respiratory Insufficiency; Postoperative Complications | interventions — Airway Extubation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Extubation in operative room: Patients are extubated in operative room after the end of surgery
  Interventions: Procedure: Extubation in operative room
- Extubation in post anesthesia care unit: Patients are extubated in post anesthesia care unit, after transfer from operative room
  Interventions: Procedure: Extubation in post anesthesia care unit

INTERVENTIONS:
Procedure: Extubation in operative room — Extubation takes place in operative room
  Groups: Extubation in operative room
Procedure: Extubation in post anesthesia care unit — Extubation takes place in post anesthesia care unit
  Groups: Extubation in post anesthesia care unit

SUMMARY:
The additional time required to awaken a patient is one of the main reasons for not extubating him or her in the operating room (OR). Conversely, transferring an intubated patient to recovery room (RR), prolonging the duration of anesthesia and intubation, in a limited environment in human resources, may lead to increased complications' rates. Little is known about those time lengths and complications rates.

DETAILED DESCRIPTION:
The additional time required to awaken a patient is one of the main reasons for not extubating him or her in the operating room (OR). Conversely, transferring an intubated patient to recovery room (RR), prolonging the duration of anesthesia and intubation, in a limited environment in human resources, may lead to increased complications' rates. Little is known about those time lengths and complications rates. The primary objective was to evaluate the additional OR occupancy time associated with awakening and extubation. Secondary objectives were to assess the rate of post-extubation complications and the need for ventilatory support. This was a prospective multicenter observational study involving intubated patients who underwent surgeries in the operating theatres of the Montpellier and Clermont-Ferrand university hospitals. Anesthesia teams were asked to complete a form including data related to the patient, surgical procedure, anesthesia procedure (induction and recovery) and the occurrence of any complications during the procedure. A multivariate analysis was conducted on the full cohort, using a propensity score (IPTW, inverse probability of treatment weighting) to account for imbalances between groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult (older than 18 years old)
* Patients admitted to any operative room of participating centre for a surgical or endoscopic procedure under general anaesthesia requiring endo-tracheal intubation
* Subjects must be covered by public health insurance
* Written informed consent from the patient or proxy (if present) before inclusion or once possible when patient has been included in a context of emergency.

Exclusion Criteria:

* Patient extubated in intensive care unit
* Patient extubated during on-call hours (because of a reduced number of medical and paramedical staff)
* Patient extubated following cardiac surgery
* Refusal of study participation or to pursue the study by the patient
* Absence of coverage by the French statutory healthcare insurance system
* Protected person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient requiring endotracheal extubation after general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 756 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Additional operative room occupancy time associated with awakening and extubation | From end of procedure until extubation, assessed up to 2 hours
  Time between dressing application (or end of procedure if there was no cutaneous effraction) and discharge from the OR

SECONDARY OUTCOMES:
Time from the end of the surgical procedure (closure of surgical site and dressing placement) to extubation | From end of procedure until extubation, assessed up to 2 hours
  Time from the end of the surgical procedure (closure of surgical site and dressing placement) to extubation
Time from the end of anaesthesia drug administration to extubation | From end of anesthesia drug administration until extubation, assessed up to 2 hours
  Time from the end of anaesthesia drug administration to extubation
Time from the end of the surgical procedure to patient able to be transferred to the ward (as defined by an Aldrete score above 10) | From end of procedure until discharge to surgical ward, assessed up to 6 hours
  Time from the end of the surgical procedure to patient able to be transferred to the ward (as defined by an Aldrete score above or equal to 10). Aldrete's scoring system is a commonly used scale for determining when postsurgical patients can be safely discharged from the post-anesthesia care unit (PACU), generally to an hospital ward, or home. Modified Aldrete score ranges from 0 to 12.
Impact of sequencing of operating programme in the room concerned on extubation location | From end of procedure until next procedure in the same room, assessed up to one day
  Impact of sequencing of operating programme in the room concerned on extubation location
Incidence of oxygen support requirement_Day-1 | First postoperative day
  Oxygen support requirement on the first day post-extubation
Reported post-operative pulmonary complications_Day7 | Seven first postoperative days
  Reported post-operative pulmonary complications within the first 7 days after extubation (as defined as acute respiratory failure, atelectasis, pneumonia, bronchospasm, pulmonary embolism or cardiorespiratory arrest)
Oxygen therapy_PACU | From end of procedure until discharge to surgical ward, assessed up to 6 hours
  Use of any rescue oxygen therapy after extubation in post-anesthesia care unit
Hypotension_PACU | From end of procedure until discharge to surgical ward, assessed up to 6 hours
  Hypotension occurrence (as defined by a systolic blood pressure below 90 mmHg and/or a mean arterial pressure below 65 mmHg)
Bradycardia_PACU | From end of procedure until discharge to surgical ward, assessed up to 6 hours
  Bradycardia occurrence (as defined as a drop of cardiac frequency below 50 beats.min-1)
Hypoxemia_PACU | From end of procedure until discharge to surgical ward, assessed up to 6 hours
  Desaturation occurrence defined as a drop of SpO2 below 96% (15), either early (within 5 min post-extubation) or delayed
NMBA_PACU | From end of procedure until discharge to surgical ward, assessed up to 6 hours
  Presence of residual neuromuscular blockade as illustrated by train of four below 90%
Reversal_NMBA | From end of anesthesia until extubation, assessed up to 2 hours
  Incidence of pharmacologic reversal of neuromuscular blocking agents
Loco-regional anaesthetic technique | Perioperative
  Use of any loco-regional anaesthetic technique
Drugs_neuromuscular blocking agents | Perioperative
  Use of neuromuscular blocking agents during anesthesia
Drugs_opioids | Perioperative
  Use of opioids during anesthesia
Drugs_hypnotics | Perioperative
  Use of hypnotics during anesthesia
Drugs_adjuvant analgesics | Perioperative
  Use of adjuvant analgesics during anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Godet, MD, PhD, Principal Investigator — Clermont-Ferrand University Hospitals; Audrey De Jong, MD, PhD, Principal Investigator — Montpellier University Hospitals
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: Undecided
Available upon reasonable request after evaluation of research question